CLINICAL TRIAL: NCT01483053
Title: A Randomised Trial Investigating the Cardiovascular Effects of Agomelatine and Escitalopram in Patients With Major Depressive Disorder.
Brief Title: Cardiovascular Effects of Agomelatine and Escitalopram in Patients With Major Depressive Disorder (MDD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baker Heart and Diabetes Institute (Other)
Collaborators: Servier Laboratories (Australia) Pty Ltd (Unknown); The Alfred (Other); Monash Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 498/11
Record Dates: First submitted 2011-11-27; First posted 2011-12-01 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major depressive disorder; Sympathetic nervous system activation; Cardiovascular risk factors; Agomelatine; Escitalopram
MeSH Terms: conditions — Depressive Disorder, Major | interventions — agomelatine; Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Agomelatine (Active Comparator): Participants who are randomly assigned to the agomelatine group will be treated with agomelatine oral tablets for twelve weeks. Participants will begin their agomelatine treatment at 25mg/day dosage, increasing to 50mg/day as clinically indicated.
  Interventions: Drug: Agomelatine
- Escitalopram (Active Comparator): Participants who are randomly assigned to the escitalopram group will be treated with escitalopram oral tablets for twelve weeks. Participants will begin their escitalopram treatment at 10mg/day dosage, increasing to 20mg/day as clinically indicated.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Agomelatine — Participants who are randomly assigned to the agomelatine group will be treated with agomelatine oral tablets for twelve weeks. Participants will begin their agomelatine treatment at 25mg/day dosage, increasing to 50mg/day as clinically indicated.
  Other Names: Valdoxan
  Arms: Agomelatine
Drug: Escitalopram — Participants who are randomly assigned to the escitalopram group will be treated with escitalopram oral tablets for twelve weeks. Participants will begin their escitalopram treatment at 10mg/day dosage, increasing to 20mg/day as clinically indicated.
  Other Names: Lexapro; Various generics, for example:; Esitalo; Esipram; Escicor; Lexam; Loxalate
  Arms: Escitalopram

SUMMARY:
There is strong evidence that patients with major depressive disorder (MDD) are at increased risk of developing coronary heart disease (CHD). This elevated risk is independent of classical risk factors such as smoking, obesity, hypercholesterolemia, diabetes and hypertension. The risk of CHD is increased 1½-2 fold in those with minor depression and 3-4½ fold in subjects with MDD. Put simply, the relative risk of developing CHD is proportional to the severity of the depression. While the mechanism of increased cardiac risk attributable to MDD is not known disturbances in autonomic function most likely do play a part.

In untreated patients with MDD (with no underlying CHD) the investigators have identified that a marked sympathetic nervous activation and diminished heart rate variability (HRV) occurs in a proportion (approximately one third) of patients. Diminished HRV has been linked to increased incidence rates of acute cardiac events in conditions such as hypertension, diabetes and myocardial infarction. Importantly, whether treating depression actually improves the risk of: (1) CHD development or (2) recurrence of cardiac events in patients with existing CHD remains unknown.

The investigators, and others, have provided a growing body of evidence linking elevated sympathetic activity and exaggerated sympathetic responses to stress to early stages of end organ dysfunction and markers of disease development. Of particular note, in addition to possible effects on HRV is the association of chronic sympathetic nervous activation to: (a) abnormal blood pressure regulation and (b) the development of insulin resistance.

The investigators therefore plan to examine the cardiovascular effects of two different antidepressant medications, agomelatine and escitalopram, in patients with MDD. In addition, the investigators plan to investigate the effects these two medications have on sympathetic nervous system activity, blood pressure, HRV, endothelial function, metabolic and psychological effects.

Findings from this study will assist us to identify of biological correlates of sympathetic nervous activation which will enable us to: (1) identify those at potentially increased cardiac risk, and (2) potentially implement additional therapeutic strategies in order to reduce cardiac risk. Indeed, it is not known whether antidepressant treatment alone would be sufficient to reverse any adverse effects of sympathetic nervous activation. This study aims to answer this important clinical question.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years.
* Capable of understanding and willing to provide signed and dated written, voluntary informed consent in advance of any protocol-specific procedures.
* MDD or MDD with melancholia according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria. Patients with comorbid panic or anxiety disorders will be included if MDD is the primary diagnosis.
* Hamilton Depression (HAM D) > 18.
* Beck Depression Inventory (BDI-II) >18.

Exclusion Criteria:

* Aged < 18 or > 65 years.
* Current antidepressant treatment.
* Previous failed response to SSRI treatment at the maximum tolerated dose for at least 4 weeks.
* Known or suspected hypersensitivity to either escitalopram or agomelatine or any of their ingredients.
* Current high suicide risk.
* Comorbid panic or anxiety disorders as the primary diagnosis.
* Pre-existing and/or current diagnosed heart disease.
* Comorbid medical conditions including type 1 diabetes, hepatic impairment (cirrhosis or active liver disease), medicated hypertension, epilepsy, bleeding disorders, alcohol/drug dependence, infectious blood diseases, psychotic disorders, personality disorders, eating disorders, mental retardation, dementia (ie, Mini Mental State Examination [MMSE] < 23), or gastrointestinal illness or previous bariatric (weight loss) surgery that may impair antidepressant absorption.
* Participants on betablockers (for example, metoprolol).
* Participants currently taking the following contraindicated medications for agomelatine and/or escitalopram:

  * Cytochrome (CYP) P450 1A2 inhibitors (e.g. fluvoxamine, ciprofloxacin)
  * Monoamine Oxidase Inhibitors;

    * Irreversible non-selective monoamine oxidase inhibitors (MAOIs)
    * Reversible, selective MAO-A inhibitor (e.g. moclobemide)
    * Reversible, non-selective MAOI (e.g. linezolid)
  * Pimozide

Participants who are eligible to take part in the study are prohibited to take the contraindicated medications listed above for the entire duration of the study.

* Clinically significant abnormalities on examination or laboratory testing and clinically significant medical conditions not listed above that are serious and/or unstable.
* Pregnant or breastfeeding women.
* Women of childbearing potential (WOCP) who are not using medically accepted contraception (ie, intrauterine devices [IUDs], hormonal contraceptives [oral, depot, patch or injectable], and double barrier methods such as condoms or diaphragms with spermicidal gel or foam). Women who are postmenopausal (ie, amenorrhea for at least 12 consecutive months) or surgically sterile are not considered to be WOCP.
* Sexually active men with WOCP partners who are not using medically accepted contraception.

Medically accepted contraception for women and sexually active men with WOCP partners will be continued throughout the study and for 30 days after the last antidepressant dose.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in markers of sympathetic nervous system activity. | Baseline and following 12 weeks of antidepressant treatment.
  The investigators will measure sympathetic nervous system activity via whole body noradrenaline spillover and microneurography. Data will be used to examine the relationship between the degree of sympathetic nervous system activity and early signs of cardiac structure and function abnormalities, insulin resistance, and morning surge in blood pressure. This may help in identifying MDD patients who are at an increased risk.

SECONDARY OUTCOMES:
Change from baseline in the magnitude of morning surge in blood pressure. | Baseline and following 12 weeks of antidepressant treatment.
  The investigators will explore the association between sympathetic nervous system activity and stress reactivity to the morning surge in blood pressure in patients with MDD. Blood pressure data will be used to test the hypothesis that MDD patients with high sympathetic activity have greater morning surges in blood pressure than patients with normal sympathetic activity.
To determine the association between sympathetic nervous system activity and left ventricular hypertrophy. | Baseline
  The investigators will measure the relationship between sympathetic nervous system activity and left ventricular mass in patients with MDD. ECG, ECHO and blood pressure data will be used to test the hypothesis that MDD patients with elevated sympathetic activity display early signs of LVH and diastolic dysfunction.
Change from baseline in insulin resistance. | Baseline and following 12 weeks of antidepressant treatment.
  The investigators will explore the association between sympathetic nervous system activity and stress reactivity to signs of insulin resistance in patients with MDD. Oral glucose tolerance data will be used to test the hypothesis that MDD patients with elevated sympathetic activity display early signs of insulin resistance.
Change from baseline on markers of cardiac risk. | Baseline and following 12 weeks of antidepressant treatment.
  The investigators will explore the association between agomelatine/escitalopram treatment and markers of cardiac risk. They will test the hypothesis that agomelatine/escitalopram treatment has a favourable effect on blood pressure variability and morning surge in blood pressure, sympathetic stress reactivity and markers of insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Lambert, Study Director — Baker IDI Heart & Diabetes Institute; David Barton, Principal Investigator — Monash Medical Centre
Locations (3):
- Australia (3):
  - Monash Medical Centre - Monash Health, Clayton, Victoria
  - Alfred and Baker Medical Unit - Alfred Hospital, Melbourne, Victoria
  - Baker IDI Heart & Diabetes Institute, Melbourne, Victoria